CLINICAL TRIAL: NCT04768595
Title: A Nutritional, Placebo Controlled, Randomised, Blinded Study of the Effect of Different Fish Oils on Omega-3 Index (CetoIndex)
Brief Title: Study of the Effect of Different Fish Oils on Omega-3 Index (CetoIndex)
Acronym: CetoIndex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Epax Norway AS (Industry)
Collaborators: Møreforsking AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: P2008
Record Dates: First submitted 2021-02-18; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Fish oil or placebo are given as gelatin capsules packaged in identical white bottles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 1g corn oil capsules
  Interventions: Dietary Supplement: Placebo
- Ceto 10 (Experimental): 1g capsules containing oil from north atlantic fish containing broad spectrum marine oil.
  Interventions: Dietary Supplement: Ceto 10
- Omega-3 (Active Comparator): 1 g capsules containing traditional, commericially available omega-3 marine oil.
  Interventions: Dietary Supplement: Fish oil

INTERVENTIONS:
Dietary Supplement: Placebo — Two, 1g capsules taken daily with food
  Arms: Placebo
Dietary Supplement: Ceto 10 — Two, 1g capsules daily with food
  Arms: Ceto 10
Dietary Supplement: Fish oil — Two, 1g capsules daily with food
  Arms: Omega-3

SUMMARY:
The study determines the EPA DHA uptake from different omega-3 supplements against a control.

DETAILED DESCRIPTION:
The chronic uptake of omega-3 fatty acids EPA and DHA are commonly determined by measurement of EPA and DHA in red bloods cells and presented as a % of total fatty acids, the so-called Omega-3 Index. The index is a validated risk assessment for cardiovascular disease. Different fish oils may influence the Omega-3 Index differently depending on their composition. This study assesses omega-3 commonly found as a supplement vs a fish oil based on north atlantic fish species.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, ≥18 -65 years of age.
2. Willing to refrain from taking omega-3 supplements for 1 month prior to study start
3. Willing to take study supplement for 2 months

Exclusion Criteria:

1. Subjects with known allergy to fish products
2. Subjects known to be pregnant or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-03-03 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Omega-3 index | Baseline (supplementation start: time point 0) to 2 months of supplementation
  Change in the omega-3 index (EPA and DHA content as a % of total fatty acids in red blood cells) from baseline to end of supplementation

SECONDARY OUTCOMES:
Change in fatty acid profile from baseline to end of supplementation between study arms. | Baseline to 2 months of supplementation.
  The secondary endpoint measures the fatty acid profiles from baseline to end of supplementation for each study arm. The results will then be compared between groups. Fatty acid profiles will be analyzed on whole blood samples using the Omega-quant test kit and analysis service. Changes in the analyzed fatty acids are determined from statistical assessment of whole blood analysis. The fatty acid profile is an exploratory endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Midtbø, PhD, Principal Investigator — Møreforsking AS
Locations (1):
- Møreforsking AS, Ålesund, Norway

IPD SHARING:
Plan to Share IPD: No